CLINICAL TRIAL: NCT04926805
Title: Physiological Study to Compare Noninvasive Ventilation (NIV) Masks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extremely slow recruitment
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIA-279; U1111-1259-4797 (Registry Identifier: WHO Universal trial number)
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Sleep-disordered Breathing; Hypercapnia
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypercapnia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mask A (Experimental): Overnight CPAP using the participant's usual pressure settings and using Mask A. One night only.
  Interventions: Device: CPAP with Mask A
- Mask B (Active Comparator): Overnight CPAP using the participant's usual pressure settings and using Mask B. One night only.
  Interventions: Device: CPAP with Mask B

INTERVENTIONS:
Device: CPAP with Mask A — CPAP mask
  Arms: Mask A
Device: CPAP with Mask B — CPAP mask
  Arms: Mask B

SUMMARY:
Noninvasive ventilation (NIV) is an established therapy that delivers positive pressure to the upper airways to provide respiratory support. Two types of NIV can be delivered; continuous positive airway pressure (CPAP) at one continuous pressure and bilevel NIV at two pressures for inhalation and exhalation.

This investigation is designed to physiologically evaluate the performance of a NIV mask, Mask A, compared to a standard NIV mask, Mask B on CPAP therapy.

People with sleep disordered breathing who have chronic hypercapnia, and are already receiving nocturnal CPAP will be recruited. They will receive one night's CPAP therapy on Mask A and 1 night on Mask B in random order. Physiological parameters will be recorded.

Parameters will be recorded during three baselines at the beginning of each evening and throughout the night when participants are asleep. The three baselines are:

1. participant awake with normal breathing (not on CPAP),
2. participant awake and on CPAP, and
3. participant asleep on CPAP in REM-sleep (rapid eye movement sleep).

ELIGIBILITY:
Inclusion Criteria:

* Already using overnight CPAP and tolerating the therapy well (over 4 hours use/night)
* Hypercapnia: venous bicarbonate of 30 milliequivalents of solute per liter (Eq/L) or more, OR transcutaneous carbon dioxide (TcCO2) of 50 millimeters of mercury (mmHg) of more.
* Provide written informed consent
* Already use a full (oronasal) face mask for CPAP
* Willing to have a venous blood sample taken during the pre-screening visit.

Exclusion Criteria:

* Presence of sleep apnea on CPAP:

  * Subjects excluded if they have an apnea-hypopnea index (AHI) of more than 20, or
  * If the AHI has not already decreased by 50 percent or more from pre-CPAP to with CPAP.
* Forced expiratory volume in 1 second (FEV1) of less than 40 percent of predicted.
* Forced expiratory volume in 1 second divided by forced vital capacity (FEV1/FVC) less than fifty percent of predicted, at the screening visit.

  * Have poorly controlled asthma or changing asthma symptoms.
  * Nasal obstruction
  * Do not fit Mask A or Mask B
  * Agitation or psychological illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Transcutaneous carbon dioxide | 1 day (From baseline to the end of the study night)
  The change in transcutaneous carbon dioxide from the 3 different baselines to the transcutaneous carbon dioxide during non-REM sleep on CPAP on the same study night. Three different values will be determined for each mask.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Veale, Dr, Principal Investigator — New Zealand Respiratory and Sleep Insitute
Locations (1):
- New Zealand Respiratory and Sleep Institute, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No